CLINICAL TRIAL: NCT05429424
Title: Complementary Acupuncture Treatment of Dysphagia in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH111-REC1-065
Record Dates: First submitted 2022-06-12; First posted 2022-06-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Stroke
Keywords: acupuncture; swallowing impairment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, the participants, assessor, and statistician are all blinded to the treatment assignments except for the acupuncturist and study coordinator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verum acupuncture group (Experimental): The study uses manual acupuncture as verum intervention.
  Interventions: Other: Verum acupuncture group
- Sham control group I (Sham Comparator): The study used specific made needle with a blunt tip, Streitberger device, as sham intervention.
  Interventions: Other: Sham control group I
- Sham control group II (Sham Comparator): Manual acupuncture at the points unrelated to the dysphagia is another sham intervention in this study.
  Interventions: Other: Sham control group II

INTERVENTIONS:
Other: Verum acupuncture group — The acupuncturist disinfected the skin of the selected acupoints with alcohol, then vertically penetrated the skin with disposable stainless-steel needles (size, brand, Taiwan) to the depth predetermined for each point (between 8-25 mm, depending on the location of the acupoint) and achieved a "deqi" response, often described as a pressure, fullness, or achiness feeling around the acupoints.
  Arms: Verum acupuncture group
Other: Sham control group I — The needle does not penetrate the skin and retract in the handle while the acupuncturist needling into the skin. The participants easily believe their intervention owing to the sensation of needling into the skin that the device mimics. The needles were fixed with a plastic ring and micropore on the body of the participants without manipulation.
  Arms: Sham control group I
Other: Sham control group II — The acupuncturist disinfected the skin of the selected acupoints with alcohol, then vertically penetrated the skin with disposable stainless-steel needles (size, brand, Taiwan) to the depth predetermined for each point (between 8-25 mm, depending on the location of the acupoint) and achieved a "deqi" response, often described as a pressure, fullness, or achiness feeling around the acupoints.
  Arms: Sham control group II

SUMMARY:
A Taiwanese study pointed out that stroke patients who have language barriers, dysphagia, and aspiration pneumonia are more likely to suffer from prolonged hospitalization. Improvements in dysphagia and subsequent complications in patients should be effective in reducing hospital stays and improving the quality of long-term care. In view of clinical medical needs and policy trends, this study aims to explore the efficacy of using traditional Chinese medicine to treat cerebral apoplexy sequelae in Taiwan. It is expected that through (1) exploration of real-world data analysis, combined with the advantages of Taiwan's biomedical database, data exploration will be carried out to provide big data (2) Multi-center prospective randomized clinical trials, providing clinical evidence of the highest level of evidence in empirical medicine.

ELIGIBILITY:
Inclusion Criteria:

* .Patients aged more than 20 years
* The diagnosis of first stroke was established within the six months
* Patients had a score ≥ 25 of Mini-Mental State Examination (MMSE)
* Patients met one or both indications as follows

  1. Dysphagia confirmed under the standardized swallowing assessment
  2. Nasogastric tube feeding already

Exclusion Criteria:

* Previous history of swallowing disability
* Currently known coagulopathy leading to bleeding disorder.
* Previous surgery of head or neck
* Local infection at or near the acupuncture site is not suitable for acupuncture after physician examination.
* Psychological or behavior disorder
* Currently pregnant or breastfeeding women.
* Previous acupuncture treatment for any indication within 30 days of enrollment.
* Severe chronic or uncontrollable complications interference the processing of the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
dysphagia severity rating scale (DSRS) | baseline, the 2nd week of the intervention, 1st and 4th week of follow-up period
  dysphagia severity rating scale(DSRS) indicates the feeding status of the dysphagia patient in three subdomains: fluids, diet, and level of supervision required for feeding. The total score from 0 to 12. The higher scores means the better outcome.
  Changes from baseline to the 2nd week of the intervention, the 1st and 4th week of follow-up period.
the functional oral intake scale (FOIS) | baseline, the 2nd week of the intervention, 1st and 4th week of follow-up period
  the functional oral intake scale(FOIS) is used to assessing the functional level of oral intake of food and liquid in stroke patients. It is a 7-point scale, with level 1 indicating complete impairment of oral intake, and level 7 indicating complete oral intake regardless of food consistency or type.
  Changes from baseline to the 2nd week of the intervention, the 1st and 4th week of follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: China Medicine University China Medicine University, Study Chair — China Medicine University
Locations (1):
- China Medical University Hospital, Taichung, Taiwan